CLINICAL TRIAL: NCT05617274
Title: Retrospective Digital Study of Mandibular Flexure in Patients With Long-span Fixed Restorations Supported by Natural Teeth.
Brief Title: Digital Assessment of Mandibular Flexure in Full Arch Fixed Restorations
Status: Completed | Type: Observational
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Medhat Sameh Abdelaziz, Principal Investigator, Future University in Egypt
Other Study IDs: FUE.REC(26)/10-2022
Record Dates: First submitted 2022-11-04; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Mandibular Flexure; Full Arch Fixed Prosthesis
Keywords: Mandibular flexure; Prosthesis Failure; Full arch restorations
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mandibular flexure before sectioning of full arch fixed prosthesis
- Mandibular flexure after sectioning of full arch fixed prosthesis
  Interventions: Procedure: Sectioning of the full arch mandibular fixed prosthesis

INTERVENTIONS:
Procedure: Sectioning of the full arch mandibular fixed prosthesis — The one unit full arch fixed prosthesis is sectioned at the midline into two pieces
  Groups: Mandibular flexure after sectioning of full arch fixed prosthesis

SUMMARY:
Nine patients (five males and four females) were included in this study who had long-term (10-15 years) of long-span rigid mandibular fixed prostheses that may have led to radiographic changes around the supporting teeth. The treatment plans included the removal of the long-span fixed rigid prostheses followed by restoring the patients with segmented implant-supported prostheses. In order to digitally measure the mandibular flexure, reference markers were adhered to the prostheses, and intraoral scans were obtained before and after splitting the preexisting prostheses at the minimum and maximum mouth opening. The distances between the markers were measured, and mandibular flexure was calculated by subtracting the distance between the markers during the maximum mouth opening from the minimum mouth opening. An independent sample T-test was used to compare mandibular flexure before and after splitting the long-span fixed prostheses.

ELIGIBILITY:
Inclusion Criteria:

* full-arch mandibular single fixed prostheses that served for many years (average 12 years) opposed by natural dentition.
* Patients were free from any systemic or debilitating diseases such as bone diseases, diabetes melilites, or blood dyscrasias.

Exclusion Criteria:

* patients with healthy fixed full-arch prosthesis
* patients with segmented prosthesis
* patients with systematic debilitating diseases.
* Patients with temporomandibular joint dysfunction, maxillofacial surgeries, or mandibular trauma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All had the entire mandibular natural dentition (6-8 abutments) splinted with a single-unit metal-ceramic (long-span fixed prosthesis). All of them suffered from different negative consequences of their one-piece fixed restorations. The retrospective collection of the patient's data was tabulated and analyzed. Nine patients were included in this study. Five males and four females, with an age range of 50-76 years were enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
change in mandibular flexure | immediately after the splitting of the full arch fixed prosthesis.
  change in mandibular flexure before and after splitting of the fixed full arch prosthesis

CONTACTS AND LOCATIONS:
Locations (1):
- Future University in Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study protocol, raw data,statistics
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] El Charkawi H, Nassar HI, Abdelaziz MS. Retrospective digital study of mandibular flexure in patients with long-span fixed restorations supported by natural teeth. BMC Res Notes. 2023 Sep 11;16(1):203. doi: 10.1186/s13104-023-06486-w. PMID 37697386